CLINICAL TRIAL: NCT02998242
Title: Apatinib in Combination With SBRT Treatment for Symptomatic Metastatic
Brief Title: Apatinib in Combination With Stereotactic Body Radiation Therapy (SBRT) Treatment for Symptomatic Metastatic Prostate Cancer
Acronym: ARCAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sichuan Provincial People's Hospital (Other)
Collaborators: Chang'An Hospital (Other); Hainan Medical College (Other)
Responsible Party: Principal Investigator, ming zeng, MD, Director of Cancer Center, Sichuan Provincial People's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ARCAP
Record Dates: First submitted 2016-12-12; First posted 2016-12-20 (Estimated); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Quality of Life
MeSH Terms: interventions — apatinib

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RT alone (Active Comparator): symptomatic bony metastatic site(s) receive SBRT less than 5 fractions
  Interventions: Radiation: SBRT to symptomatic bony metastatic bony site(s)
- RT with apatinib (Experimental): selected dose administered PO during and after SBRT
  Interventions: Drug: Apatinib; Radiation: SBRT to symptomatic bony metastatic bony site(s)

INTERVENTIONS:
Drug: Apatinib
  Arms: RT with apatinib
Radiation: SBRT to symptomatic bony metastatic bony site(s)

SUMMARY:
To study safety and efficacy of apatinib in combination of radiotherapy in patients with symptomatic bony disease prostate cancer (SBPC), based on the potential synergistic antitumor activity between Apatinib and Stereotactic Body Radiation Therapy (SBRT).

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of adenocarcinoma of the prostate
* Metastatic and symptomatic prostate cancer (positive bone scan or measurable disease)
* Patients must stop using any herbal product known to decrease PSA levels (eg., saw palmetto and PC-SPES) or any systemic or topical corticosteroid at least 4 weeks prior to screening. Progressive disease must be documented after discontinuation of these products.
* Progressive disease after androgen deprivation (or hormone therapy). For patients with measurable disease, progression will be defined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria. For patients with progression in, or without any measurable disease, a positive bone scan and elevated PSA will be required.
* Patients receiving bisphosphate therapy must have been on stable doses for at least 4 weeks with stable symptoms prior to enrollment.
* No prior chemotherapy or immunotherapy (tumor vaccine, cytokine, or growth factor given to control prostate cancer).
* Prior radiation therapy completed at least 4 weeks prior to enrollment. No prior radiopharmaceuticals (strontium, samarium) within 8 weeks prior to enrollment.

Exclusion Criteria:

* History of severe hypersensitivity reactions to drugs formulated with polysorbate 80.
* Patients with active autoimmune disease or a history of autoimmune disease that required systemic steroids or immunosuppressive medications, except for patients with vitiligo.
* Prior therapy with any anti-cytotoxic T-lymphocyte antigen 4 (anti-CTLA-4) antibody.
* Active infection requiring therapy.
* Concurrent medical condition requiring the use of systemic or topical corticosteroids; systemic or topical corticosteroids must be discontinued at least 4 weeks prior to enrollment. The use of inhaled corticosteroids is acceptable.

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-05-10 (Actual); Primary Completion 2017-01-05 (Actual); Study Completion 2017-12-10 (Actual)

PRIMARY OUTCOMES:
biochemical disease free survival | 2 years

IPD SHARING:
Plan to Share IPD: Yes